CLINICAL TRIAL: NCT06939283
Title: A Phase 1b/2 Multisite Dose- and Regimen-finding and Expansion Study of WTX-330 in Adult Patients With Selected Advanced or Metastatic Solid Tumors or Non-Hodgkin Lymphoma (NHL)
Brief Title: A Phase 1b/2 Multisite Dose-finding and Expansion Study of WTX-330 in Adult Patients With Selected Advanced or Metastatic Solid Tumors or Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Werewolf Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WTX-330x2102
Record Dates: First submitted 2025-03-26; First posted 2025-04-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Advanced or Metastatic Solid Tumors; Non-Hodgkin Lymphoma
Keywords: WTX-330; Cancer; Immunotherapy; Interleukin-12; IL-12; Checkpoint inhibitor resistance
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose- and Regimen Finding (Experimental): Regimen 1 Fixed Dose for 28 days then Regimen 2 Step-up Dose for 28 days
  Interventions: Drug: WTX-330
- Dose Expansion Arm A (Experimental): n~20 Patients with locally advanced or metastatic cutaneous malignant melanoma who have been treated with a standard of care (SOC) checkpoint inhibitor (CPI) regimen and who demonstrate primary or secondary resistance to this therapy
  Interventions: Drug: WTX-330
- Dose Expansion Arm B (Experimental): n~20 Patients with locally advanced or metastatic microsatellite-stable (MSS) colorectal carcinoma (CRC) who have progressed on or are intolerant of SOC therapies and who are naïve to immunotherapy
  Interventions: Drug: WTX-330
- Dose Expansion Arm C (Experimental): n~20 Patients with advanced NHL who are relapsed/refractory to SOC therapies and who are CPI naïve
  Interventions: Drug: WTX-330

INTERVENTIONS:
Drug: WTX-330 — Investigational Product

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of the study drug WTX-330 when administered using a fixed dose regimen or a step-up dose regimen in adult patients with selected advanced or metastatic solid tumors or lymphoma. In addition to safety and tolerability, the study aims to:

* determine the maximum initial dose of WTX-330 that may be used in the step-up dose regimen
* determine whether the step-up dose regimen can increase WTX-330 exposure in patients due to improved tolerability
* determine the maximum tolerated dose (MTD) of WTX-330 and/or recommended dose for expansion (RDE) for each regimen
* evaluate the antitumor activity of WTX-330
* characterize the pharmacokinetic (PK) profile of WTX-330
* characterize the interferon gamma (IFNγ) profile after treatment with WTX-330
* evaluate changes in immunological biomarkers
* determine the impact of WTX-330 on overall survival (OS)

Study participants will participate in a dose- and regimen-finding phase (Part 1) followed by a dose expansion phase (Part 2) where they will be assigned to one of three arms (A, B and C).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Dose escalation (Part 1): Patients with relapsed/refractory locally advanced or metastatic solid tumor for which the patient has progressed on or is intolerant of standard therapy, or for whom no standard therapy with proven benefit exists. Patients with castrate resistant prostate cancer (CRPC) and primary Central Nervous System (CNS) malignancies are ineligible. Patients with non-Hodgkin lymphoma (NHL) will not be enrolled in the dose escalation but are eligible for the dose expansion.
3. Dose Expansion (Part 2): Patients with relapsed/refractory locally advanced or metastatic cutaneous melanoma, MSS CRC or NHL for which the patient has progressed on or is intolerant of standard therapy. The dose expansion consists of 3 arms (A, B and C) with the following eligibility criteria:

   * Arm A: Patients with locally advanced or metastatic cutaneous melanoma who demonstrate either primary or secondary resistance to checkpoint inhibitor (CPI) therapy. Patients must have received at least 1 prior line that was a SOC CPI regimen and are allowed no more than 3 prior lines for advanced disease. Prior T-VEC therapy is allowed and does not count as a prior line, but treated lesions cannot be used as target lesions or accessed for mandatory pre- and on-treatment biopsies.
   * Arm B: Patients with relapsed/refractory locally advanced or metastatic MSS CRC who are immunotherapy naïve. Patients should have had no more than 3 prior lines of therapy in the advanced/metastatic setting and must have either progressed on or be intolerant of the certain agents.
   * Arm C: Patients with advanced NHL who have follicular lymphoma or diffuse large B-cell lymphoma (DLBCL). Other subtypes of NHL may be considered after discussion with the Sponsor. All patients with NHL must have received at least 2 prior systemic therapies and have relapsed or refractory disease. Prior therapy with autologous Chimeric Antigen Receptor T-Cell (CAR-T) therapy is permitted and will be considered a prior line.
   * Patients with follicular lymphoma (or other indolent lymphoma)
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. At least one measurable lesion per RECIST 1.1 or evaluable lesion per Lugano classification.
6. Agrees to undergo a pre-treatment and on-treatment biopsy of a primary or metastatic tumor lesion.
7. Human immunodeficiency virus (HIV) infected patients must be on antiretroviral therapy (ART) and well-controlled HIV infection/disease
8. Has adequate organ and bone marrow function.
9. Willingness of men and women of reproductive potential to agree to highly effective birth control for the duration of treatment and for 4 months following the last dose of study drug.

Exclusion Criteria:

1. A history of another active malignancy (a second cancer) within the previous 2 years, except for localized cancers that are not related to the current cancer being treated, is considered cured, and, in the opinion of the Investigator, presents a low risk of recurrence. These exceptions include, but are not limited to, basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
2. Received prior treatment with IL-12 by any route of administration (including intratumoral injection).
3. Patients with primary CNS malignancies and CRPC
4. Have known symptomatic brain metastases requiring steroids.
5. Significant cardiovascular disease
6. Significant electrocardiogram (ECG) abnormalities
7. Active autoimmune disease requiring systemic treatment in the past 2 years
8. Diagnosis of immunodeficiency, on immunosuppressive therapy, or receiving chronic systemic or enteric steroid therapy (dose > 10 mg/day of prednisone or equivalent)
9. Major surgery (excluding placement of vascular access) within 2 weeks prior to the first dose of study drug.
10. Investigational agent or anticancer therapy (including chemotherapy, biologic therapy, immunotherapy, anticancer Chinese medicine, or other anticancer herbal remedy) within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study drug.
11. Radiotherapy within 2 weeks of start of study treatment. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
12. Any unresolved toxicities from prior therapy greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 Grade 1 at the time of starting study drug with the exception of alopecia Grade 2 platinum therapy-related neuropathy and Grade 2 endocrine immune-related AEs managed with a stable dose of hormone replacement therapy.
13. Use of sensitive substrates of major CYP450 isozymes.
14. Any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign the informed consent form (ICF), adversely affect the patient's ability to cooperate and participate in the study, or compromise the interpretation of study results.
15. Received a live vaccine within 30 days of the first dose of study drug.
16. Active systemic bacterial, viral, or fungal infection.
17. HIV-infected participants with a history of Kaposi sarcoma and/or multicentric Castleman Disease.
18. Active infection as determined by hepatitis B surface antigen and hepatitis B core antibody, or hepatitis B virus deoxyribonucleic acid (DNA) by quantitative polymerase chain reaction (qPCR) testing.
19. Active infection as determined by hepatitis C virus (HCV) antibody or HCV RNA by qPCR testing.
20. Pregnant or lactating.
21. History of hypersensitivity to any of the study drug components.
22. Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | 4 weeks
Incidence of treatment emergent adverse events | 24 months
Incidence of changes in clinical laboratory abnormalities | 24 months
Overall response rate (ORR) by response evaluation criteria in solid tumors (RECIST) 1.1 and the immune-overall response rate (iORR) by immune RECIST (iRECIST; Part 2, Arms A and B) or response by Lugano classification (Part 2, Arm C) | 24 months
Duration of response (DOR) by response evaluation criteria in solid tumors (RECIST) 1.1 and immune RECIST (iRECIST; Part 2, Arms A and B) or based on Lugano classification (Part 2, Arm C) | 24 months

SECONDARY OUTCOMES:
Characterize the plasma concentrations of WTX-330, free IL-12 and interferon gamma (IFNγ) | 24 months
Changes in PD-L1 expression in tumor biopsies | 24 months
Duration of response (DOR) by response evaluation criteria in solid tumors (RECIST) 1.1 and immune RECIST (iRECIST; Part 1 and Part 2, Arms A and B) or based on Lugano classification (Part 2, Arm C) | 24 months
Progression-free survival (PFS) by response evaluation criteria in solid tumors (RECIST) 1.1 and immune RECIST (iRECIST; Part 1 and Part 2, Arms A and B) or based on Lugano classification (Part 2, Arm C) | 24 months
Overall survival (OS) after treatment with WTX-330 in Part 2 based on death, start of new anticancer therapies, withdrawal of consent or lost to follow-up | 36 months
Incidence of WTX-330 antidrug antibodies | 24 months
Titers of WTX-330 antidrug antibodies | 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - NEXT Oncology, San Antonio, Texas